CLINICAL TRIAL: NCT03283982
Title: Registry-Based, Prospective, Single-Blind, Randomized Controlled Trial: Robotic vs. Laparoscopic Ventral Hernia Repair With Intraperitoneal Onlay Mesh (IPOM)
Brief Title: Laparoscopic vs. Robotic Ventral Hernia Repair With IPOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Principal Investigator, Ajita Prabhu, MD, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-1053
Record Dates: First submitted 2017-09-08; First posted 2017-09-15 (Actual); Results first posted 2022-07-19 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Ventral Hernia
Keywords: Ventral Hernia; Robotic; Laparoscopic; Pain scores
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Robotic IPOM (Active Comparator): Robotic Ventral Hernia Repair with IPOM: The da Vinci® Surgical System robotic platform (Intuitive Surgical, Inc.) will be used to perform a minimally invasive ventral hernia repair with intraperitoneal mesh placement.
  Interventions: Device: Robotic Ventral Hernia Repair with IPOM
- Laparoscopic IPOM (Active Comparator): Laparoscopic Ventral Hernia Repair with IPOM: The standard laparoscopic platform will be used to perform a minimally invasive ventral hernia repair with intraperitoneal mesh placement.
  Interventions: Device: Laparoscopic Ventral Hernia Repair with IPOM

INTERVENTIONS:
Device: Robotic Ventral Hernia Repair with IPOM — Minimally invasive ventral hernia repair with intraperitoneal mesh placement, using the da Vinci robotic platform
  Other Names: da Vinci® Surgical System robotic platform
  Arms: Robotic IPOM
Device: Laparoscopic Ventral Hernia Repair with IPOM — Minimally invasive ventral hernia repair with intraperitoneal mesh placement, using the laparoscopic platform
  Arms: Laparoscopic IPOM

SUMMARY:
The investigators aim to conduct a registry-based, randomized controlled trial to investigate if the robotic platform for minimally invasive ventral hernia repair with intraperitoneal onlay mesh (IPOM), when compared to the laparoscopic platform, will influence on early postoperative pain scores, wound morbidity (surgical site infections, surgical site occurrences and surgical site occurrences requiring procedural intervention), ventral hernia recurrence rate and abdominal wall-specific quality of life.

DETAILED DESCRIPTION:
Despite the adoption of the robotic platform for ventral hernia repair, there is still a paucity of literature to speak to the benefits of this approach. In a recently-published propensity score analysis comparing laparoscopic and robotic ventral hernia repairs with intraperitoneal onlay mesh (IPOM) , the authors showed a 1-day decrease in hospital length of stay (LOS) with the robotic versus laparoscopic platform for laparoscopic ventral hernia repair with IPOM. The reasons for this decrease in stay remain unknown. While multiple papers have described postoperative pain scores following laparoscopic ventral hernia repair, scant data exists evaluating postoperative pain following robotic ventral hernia repair. To help determine if the robotic platform has an impact on postoperative pain, wound morbidity rates, ventral hernia recurrence and quality of life, the investigators propose a registry-based, randomized clinical trial (RCT) through the Americas Hernia Society Quality Collaborative (AHSQC). The AHSQC is a multicenter, nationwide quality improvement effort with a mission to improve value in hernia care. Data are collected prospectively in the routine care of hernia patients for quality improvement purposes. The information collected in the AHSQC offers a natural repository of information that can be used for research, in addition to its quality improvement purpose. The investigators aim to conduct a prospective, registry-based, single-blind, randomized controlled trial with a 1:1 allocation ratio. This will be a single-institutional study performed at the Cleveland Clinic Foundation in Cleveland, Ohio from 2017 to 2020. All enrollments and surgeries in this study will take place at the Cleveland Clinic Comprehensive Hernia Center. The study will consist of 2 interventions: laparoscopic IPOM or robotic IPOM. Participants will be randomized to laparoscopic ventral hernia repair with IPOM or robotic ventral hernia repair with IPOM at the moment of enrollment, during preoperative evaluation. Participants will be blinded to the intervention. Both the laparoscopic and robotic platforms represent current standards of care for ventral hernia repair, and both approaches are currently offered at Cleveland Clinic Comprehensive Hernia Center. The sample size was determined by the primary outcome of interest, the change in NRS-11 pain score at postoperative day 1. The investigators hypothesize that the robotic approach will be associated with a 30% decrease in NRS-11 pain score at postoperative day 1. The 30% reduction used for power calculations was determined from clinical judgment, as little literature exists evaluating the minimal clinically important difference of the NRS-11 scale for ventral hernia repair. Mean NRS-11 pain score (4.76) and standard deviation (1.975) with the laparoscopic approach (control group) was determined from previously published manuscripts. Assuming an alpha of 0.05, a beta of 0.20, a total sample size of 62 patients (31 per arm) was calculated. Considering and a 20% drop-out rate to occur in each arm, approximately 74 patients (37 patients per arm) was defined as the sample size for this study. Descriptive statistics, including means, standard deviations, and/or percentages, will be calculated for demographic and baseline variables. Categorical variables will be reported using proportions. Continuous variables will be reported using either means and standard deviations for normally distributed data or median and interquartile range for non-parametric data. Pain scores will be compared between intervention arms at each time point using either a Student's t-test (normal distribution) or a Kruskal-Wallis test (nonparametric distribution). Differences in PROMIS scores between baseline, 30 and 365 days, respectively, will be assessed via Wilcoxon signed-rank test. Recurrence rates will be compared between intervention arms via Pearson's chi-square. Abdominal wall-specific quality of life scores will be compared between intervention arms via Kruskal-Wallis test. Wound events will be compared between intervention arms via Pearson's chi-square.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* Primary or Incisional Ventral Hernia
* Midline defect location
* H. Width equal or less than 7 centimeters
* Elective setting
* Able to give informed consent
* Able to tolerate general anesthesia
* Considered eligible for minimally invasive ventral hernia repair
* Willing to undergo mesh-based repair
* Fascial closure is presumed to be achieved

Exclusion Criteria:

* Younger than 18 years old
* Non-midline hernia defects
* H. Width > 7cm
* Emergent setting ( acute incarceration or strangulation)
* Unable to give informed consent
* Unable to tolerate general anesthesia
* Considered not eligible for minimally invasive ventral hernia repair
* Not willing to undergo mesh based repair
* Fascial closure not intended or presumed not to be achieved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajita Prabhu, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Comprehensive Hernia Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Background] Prabhu AS, Dickens EO, Copper CM, Mann JW, Yunis JP, Phillips S, Huang LC, Poulose BK, Rosen MJ. Laparoscopic vs Robotic Intraperitoneal Mesh Repair for Incisional Hernia: An Americas Hernia Society Quality Collaborative Analysis. J Am Coll Surg. 2017 Aug;225(2):285-293. doi: 10.1016/j.jamcollsurg.2017.04.011. Epub 2017 Apr 24. PMID 28450062
- [Background] Asencio F, Aguilo J, Peiro S, Carbo J, Ferri R, Caro F, Ahmad M. Open randomized clinical trial of laparoscopic versus open incisional hernia repair. Surg Endosc. 2009 Jul;23(7):1441-8. doi: 10.1007/s00464-008-0230-4. Epub 2008 Dec 31. PMID 19116750
- [Derived] Petro CC, Thomas JD, Tu C, Krpata DM, Beffa LR, Rosen MJ, Prabhu AS. Robotic vs Laparoscopic Ventral Hernia Repair with Intraperitoneal Mesh: 1-Year Exploratory Outcomes of the PROVE-IT Randomized Clinical Trial. J Am Coll Surg. 2022 Jun 1;234(6):1160-1165. doi: 10.1097/XCS.0000000000000171. Epub 2022 Mar 14. PMID 35703814
- [Derived] Petro CC, Zolin S, Krpata D, Alkhatib H, Tu C, Rosen MJ, Prabhu AS. Patient-Reported Outcomes of Robotic vs Laparoscopic Ventral Hernia Repair With Intraperitoneal Mesh: The PROVE-IT Randomized Clinical Trial. JAMA Surg. 2021 Jan 1;156(1):22-29. doi: 10.1001/jamasurg.2020.4569. PMID 33084881

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Robotic IPOM | Laparoscopic IPOM
Started | 39 | 36
Completed | 39 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Robotic IPOM | Laparoscopic IPOM | Total
Number analyzed (Participants) | 39 | 36 | 75
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 56 [50 to 69.5] | 55.5 [49 to 59.5] | 56 [49 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 37
  Male | 23 | 15 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black/ African American | 6 | 7 | 13
  Race: White | 33 | 29 | 62

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Scores
Description: Pain scores will be assessed using the Numeric Pain Rating Scale (NRS-11); The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"); This will be reported using median and interquartile ranges
Time Frame: Pain scores will be assessed on postoperative day 1, day 7 and day 30
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Robotic IPOM | Laparoscopic IPOM
Number analyzed (Participants) | 39 | 36
score on a scale
  Post Surgery Day 1 | 5 [3 to 6] | 5 [3 to 7]
  Post Surgery Day 7 | 4 [2 to 5] | 3 [2 to 5]
  Post Surgery Day 30 | 1 [0 to 2] | 2 [0 to 3.5]

2. Primary Outcome: Postoperative Pain Scores
Description: Pain scores will be assessed using the PROMIS (Patient-Reported Outcomes Measurement Information System) 3a Pain Intensity Survey. Measured on a scale of 30.7- 71.8 with the higher numbers indicating higher pain
Time Frame: 30 days(+-15days) postoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Robotic IPOM | Laparoscopic IPOM
Number analyzed (Participants) | 39 | 36
score on a scale | 44.9 [40.2 to 50.1] | 46.3 [40.2 to 49.4]

3. Secondary Outcome: Number of Participants With Central Hernia Recurrence
Description: Ventral Hernia recurrence will be assessed at 1 year postoperatively, either by physical examination, imaging studies or using the validated Ventral Hernia Recurrence Inventory Survey. Rates of ventral hernia recurrence will be reported as percent
Time Frame: 12 months +- 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic IPOM | Laparoscopic IPOM
Number analyzed (Participants) | 39 | 36
Participants | 2 | 1

4. Secondary Outcome: Cost of Robotic IPOM Versus Laparoscopic IPOM
Time Frame: Start of procedure to end of procedure which is an average of 2 hours
Measure: Median (Inter-Quartile Range); unit: American Dollars
Arm/Group | Robotic IPOM | Laparoscopic IPOM
Number analyzed (Participants) | 39 | 36
American Dollars | 2438 [1942 to 3245] | 2102 [1826 to 2530]

5. Other Pre Specified Outcome: Abdominal Wall Specific Quality of Life
Description: Abdominal Wall Specific Quality of Life will be assessed using the validated HerQLes (Hernia Related Quality of Life) survey. Scores will be reported as mean and standard deviations as appropriate on a scale from 0-100 with the larger numbers representing higher quality of life.
Time Frame: 30-days(+-15days) postoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Robotic IPOM | Laparoscopic IPOM
Number analyzed (Participants) | 39 | 36
score on a scale | 67 [46 to 80.8] | 72 [35 to 80]

6. Other Pre Specified Outcome: Number of Participants With Surgical Site Infection
Description: Surgical site infection rates will be assessed and reported as percent
Time Frame: 30 days +- 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic IPOM | Laparoscopic IPOM
Number analyzed (Participants) | 39 | 36
Participants | 0 | 0

7. Other Pre Specified Outcome: Number of Participants With Surgical Site Occurrences Requiring Procedural Intervention
Description: Surgical Site Occurrences requiring Procedural Intervention will be assessed and reported as percent
Time Frame: 30 days +- 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic IPOM | Laparoscopic IPOM
Number analyzed (Participants) | 39 | 36
Participants | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Surgical Site Occurrences
Description: Surgical site occurrences ( defined as wound cellulitis, non-healing wound, fascial disruption, skin or soft tissue ischemia or necrosis, wound drainage, stitch abscess, seroma, hematoma, exposed, contaminated or infected mesh and enterocutaneous fistula) will be assessed and reported as percent
Time Frame: 30-days +- 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic IPOM | Laparoscopic IPOM
Number analyzed (Participants) | 39 | 36
Participants
  None | 38 | 36
  Yes | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year post surgery
Arm/Group | Robotic IPOM | Laparoscopic IPOM
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/39 | 0/36
Other Adverse Events (participants affected / at risk) | 5/39 | 6/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic IPOM (N=39) | Laparoscopic IPOM (N=36)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic IPOM (N=39) | Laparoscopic IPOM (N=36)
Pain (General disorders) | 1 (1) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 3 (3)
Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Scar Revision (Surgical and medical procedures) | 1 (1) | 0 (0)
Access-Related Injury (Surgical and medical procedures) | 1 (1) | 0 (0) — Injury occurring during the procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT03283982/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT03283982/ICF_001.pdf